CLINICAL TRIAL: NCT01903434
Title: A Bioequivalence Study in Healthy Subjects Administered Evacetrapib Tablets of Varying Tablet Solid Fractions
Brief Title: A Study of Evacetrapib (LY2484595) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14623; I1V-MC-EIAU (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evacetrapib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evacetrapib -- Solid Fraction Test (Experimental): Single oral dose of 130 milligram (mg) evacetrapib tablet on Day 1 of up to 2 of 3 periods
  Interventions: Drug: Evacetrapib
- Evacetrapib -- Solid Fraction Reference (Experimental): Single oral dose of 130 mg evacetrapib tablet on Day 1 of up to 2 of 3 periods
  Interventions: Drug: Evacetrapib

INTERVENTIONS:
Drug: Evacetrapib — Administered orally
  Other Names: LY2484595

SUMMARY:
The purpose of this study is to measure and compare the amounts of the study drug evacetrapib found in the blood after taking two different formulations. The study has 3 periods. Participants will take each formulation by mouth at least once. A minimum of 14 days will pass between study drug doses. The safety and tolerability of the study drug will also be examined. Information about any side effects that may occur will also be collected. This study will last approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who agree to use a reliable method of birth control and not donate sperm during the study and for 90 days after study completion
* Female participants who are not of child-bearing potential due to surgical sterilization confirmed by medical history or menopause
* Have a body mass index of 18 to 32 kilograms per square meter (kg/m^2)
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Are currently enrolled in or have completed or discontinued within the last 30 days from a clinical trial involving an investigational product
* Have known allergies to evacetrapib, related compounds or any components of the formulation, or history of significant allergic disease as determined by the investigator
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Are women who are pregnant or lactating
* Have used or intend to use over-the-counter or prescription medications (including vitamins/mineral supplements, herbal medicine) 14 days prior to enrollment and during the study
* Have donated blood of more than 500 milliliters (mL) within the last month
* Have an average weekly alcohol intake that exceeds 21 units per week (for males) and 14 units per week (for females) or are unwilling to stop alcohol consumption 48 hours prior to each dose and while resident at the Clinical Research Unit (CRU)
* Currently smoke or use tobacco or nicotine products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Reference/Test/Test: A single dose of Reference 130 mg evacetrapib on Day 1 of Period 1 and of Test 130 mg evacetrapib on Day 1 of Period 2 and Day 1 of Period 3.
  There was a washout period of at least 14 days between doses. Each participant received up to 3 doses.
- Test/Reference/Reference: A single dose of Test 130 mg evacetrapib on Day 1 of Period 1 and of Reference 130 mg evacetrapib on Day 1 of Period 2 and Day 1 of Period 3.
  There was a washout period of at least 14 days between doses. Each participant received up to 3 doses.
Period: Treatment Period 1
Arm/Group | Reference/Test/Test | Test/Reference/Reference
Started | 30 | 30
Received at Least 1 Dose of Study Drug | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: Washout Period 1 (at Least 14 Days)
Arm/Group | Reference/Test/Test | Test/Reference/Reference
Started | 30 | 30
Completed | 29 | 28
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Period: Treatment Period 2
Arm/Group | Reference/Test/Test | Test/Reference/Reference
Started | 29 | 28
Received at Least 1 Dose of Study Drug | 29 | 28
Completed | 29 | 28
Not Completed | 0 | 0
Period: Washout Period 1 (at Least 14 Days)
Arm/Group | Reference/Test/Test | Test/Reference/Reference
Started | 29 | 28
Completed | 29 | 28
Not Completed | 0 | 0
Period: Treatment Period 3
Arm/Group | Reference/Test/Test | Test/Reference/Reference
Started | 29 | 28
Received at Least 1 Dose of Study Drug | 29 | 28
Completed | 29 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at last 1 dose of evacetrapib.
Groups:
- 130 mg Evacetrapib: Participants randomized to receive a single dose of 130 mg evacetrapib of either of the two different solid fraction controls on Day 1 of each of 3 treatment periods, according to their assigned treatment sequence.
Arm/Group | 130 mg Evacetrapib
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 39
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Evacetrapib (LY2484595)
Description: The maximum observed drug concentration (Cmax) of evacetrapib is summarized for each solid fraction control (Reference and Test).
Time Frame: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose in each period
Population: Participants who received at least 1 dose of evacetrapib and had evaluable evacetrapib concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Groups:
- Reference: Evacetrapib: 130 mg with a solid fraction of 0.86 administered on Day 1 of up to 2 of 3 treatment periods.
- Test: Evacetrapib: 130 mg with a solid fraction of 0.89 administered on Day 1 of up to 2 of 3 treatment periods.
Arm/Group | Reference | Test
Number analyzed (Participants) | 58 | 59
nanograms per milliliter | 604 (76) | 597 (102)

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Evacetrapib (LY2484595)
Description: Evacetrapib exposure in terms of Area Under the Concentration Versus Time Curve from time 0 extrapolated to infinity (AUC[0-∞]) is summarized for each solid fraction control (Reference and Test).
Time Frame: as for outcome 1
Population: Participants who received at least 1 dose of evacetrapib and had evaluable evacetrapib concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms times hours per milliliter
Arm/Group | Reference | Test
Number analyzed (Participants) | 58 | 59
nanograms times hours per milliliter | 10400 (56) | 10300 (68)

ADVERSE EVENTS:
Arm/Group | Reference | Test
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/59
Other Adverse Events (participants affected / at risk) | 4/58 | 1/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference (N=58) | Test (N=59)
Headache (Nervous system disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days